CLINICAL TRIAL: NCT05876871
Title: Quantitative Stress Radiography With Pelvic Binder for Evaluation of Instability in Lateral Compression Pelvic Ring Injuries
Brief Title: Stress Radiography for Pelvic Ring Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Joseph Patterson, Assistant Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-22-00217
Record Dates: First submitted 2022-09-28; First posted 2023-05-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Fracture
Keywords: pelvic binder; pelvic ring injury; pelvic instability; stress radiography
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic Intervention (Other)
  Interventions: Diagnostic Test: Pelvic Binder Radiography

INTERVENTIONS:
Diagnostic Test: Pelvic Binder Radiography — One series of radiographic exposures

SUMMARY:
The primary aim of this investigation is to prospectively and clinically validate a novel, reproducible method of quantitative application of compressive stress to a LC1 pelvic ring injury of indeterminate stability for the purpose of assessing quantitative pelvic ring displacement.

DETAILED DESCRIPTION:
patients will receive a diagnostic intervention with multiple x-rays. These x-rays will be taken as different levels of force are applied to the pelvis. This will be used to determine instability as an indication for surgical intervention to stabilize the pelvic ring.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Acute emergency department admission or transfer to Los Angeles County + USC Medical Center
* Presentation within 3 weeks of injury
* Blunt or blast mechanism of traumatic injury
* Lateral compression pelvic ring injury with unilateral incomplete disruption of the posterior arch (OTA/AO 61B1.1/2.2; Young Burgess LC1) on radiographs and/or computed tomography scan of the pelvis obtained per routine care
* LC1 pelvic ring injuries occurring in isolation are virtually never associated with hemodynamic instability or critical patient condition
* Stress examination of LC1 pelvic ring injury is standard of care
* Patient must speak either English or Spanish

Exclusion Criteria:

* Volume expanding pelvic ring injury (Young-Burgess APC-2 and 3, LC-3, vertical shear, and combined mechanism of injury (CMI) (Tile B and C patterns; OTA codes 61-B and 61-C).
* Volume expanding pelvic ring injury injuries represent the types of pelvic ring disruption responsible for pelvic hemorrhage and hypotension and are correlate with patient hemodynamic instability as well as critical injuries
* Volume expanding pelvic ring injury injuries warrant stabilization with circumferential pelvic compression.
* Patients with volume expanding pelvic ring injury are not clinically appropriate for this study.
* Hemodynamic instability or hypotension angioembolization (AE), preperitoneal pelvic packing (PPP), or Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) to obtain or maintain hemodynamic stability
* Bladder, vaginal, rectal, colonic, or other abdominal or pelvic organ injury precluding safe application of circumferential pelvic compression device
* Patient likely to have severe problems with maintaining follow- up due to at least one of the following:
* Patient has been diagnosed with a severe psychiatric condition
* Patient is intellectually challenged without adequate family support
* Patient lives outside the hospital's catchment area
* Follow-up is planned at another medical center
* Patients who are prisoners or homeless

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Pelvic fracture displacement at 5 kg of stress | At diagnostic intervention, immediately following baseline data collection.
  Linear displacement of the pelvis fracture defined as the difference in distance measured at the acetabular teardrops on a pelvis inlet radiograph with no applied stress and a pelvis inlet radiograph with 5 kg of stress applied with the pelvic binder.
Pelvic fracture displacement at 10 kg of stress | At diagnostic intervention, immediately following baseline data
  Linear displacement of the pelvis fracture defined as the difference in distance measured at the acetabular teardrops on a pelvis inlet radiograph with no applied stress and a pelvis inlet radiograph with 10 kg of stress applied with the pelvic binder.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Patterson, MD, Principal Investigator — Keck School of Medicine of the University of Southern California
Locations (1):
- Keck Medical Center of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No